CLINICAL TRIAL: NCT01193283
Title: Cyclophosphamide Plus Cyclosporine in Treatment-Naive Severe Aplastic Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Danielle Townsley, M.D., Hematology Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100176; 10-H-0176 (Other: NIH NHLBI)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Aplastic Anemia; Neutropenia; Pancytopenia; Severe Aplastic Anemia
Keywords: Aplastic Anemia; Immunosuppression; T-Cells; Hematopoiesis; Autoimmunity; Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic; Neutropenia; Pancytopenia; Autoimmune Diseases | interventions — Cyclophosphamide; Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SAA hematologic response (Experimental): Treatment-naive severe aplastic anemia patients will receive a low dose of cyclophosphamide (120mg/kg) and low dose cyclosporine ( target therapeutic level of 100-200 micrograms per liter). Cyclophosphamide will be given once daily for 4 doses. Cyclosporine will be started after cyclophosphamide completion, cyclosporine will be given twice daily. The dosing will be modified to attain the therapeutic level.
  Interventions: Drug: Cyclophosphamide; Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclophosphamide — 30 my/kg for 4 days
  Other Names: Cytoxan
Drug: Cyclosporine — daily to a trough of 100 t0 200 ng/ml
  Other Names: Gengraf; Neoral; Sandimmune

SUMMARY:
Background:

* Severe aplastic anemia (SAA) can lead to problems with bone marrow health and result in low blood cell counts, which require frequent transfusions. Standard treatment for SAA involves injections of antithymocyte globulin (ATG) plus cyclosporine (CsA). This regimen has been shown to improve the blood counts in about two-thirds of patients. However, the ATG/CsA regimen has the following limitations: (a) the disease can come back (relapse) in about one-third of patients who improve initially; and (b) in about 10% to 15% of cases, certain types of bone marrow cancer (such as myelodysplasia and leukemia) can develop (called evolution). Experience with other drugs in SAA such as cyclophosphamide suggests that similar response rates to ATG/CsA can be achieved with a lower risk of relapse and clonal evolution. However, cyclophosphamide was found to have significant side effects in SAA when investigated over 10 years ago due to increase risk of fungal infections.
* Better antibiotic drugs against fungus have been developed and are widely used to treat patients who have low white blood cell counts and are at risk of developing infections. In SAA patients in particular, these newer antibiotics have had a large impact in preventing and treating fungus infections. Researchers are revisiting the use of cyclophosphamide in SAA treatment, and plan to give a lower dose of CsA in combination with the immune-suppressing drug cyclophosphamide, as well as antibiotics to protect against infections, as a possible treatment for the disease.

Objectives:

- To determine the safety and effectiveness of the combination of cyclophosphamide and cyclosporine in treating severe aplastic anemia that has not been treated with immunosuppressive therapy.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Allogeneic hematopoietic stem cell transplantation (HSCT) offers the opportunity for cure in 70 percent of patients, but most patients are not suitable candidates for this treatment modality due to advanced age, comorbidities or lack of a histocompatible donor. For these patients, comparable long-term survival is attainable with immunosuppressive treatment (IST) with anti-thymocyte globulin (ATG) and cyclosporine (CsA). However, approximately 1/3 of patients do not show blood count improvement after ATG/CsA and are considered to have refractory disease. Furthermore, analysis of our own extensive clinical data suggests that poor blood count responses to a single course of ATG (non-robust responders), even when transfusion-independence is achieved, predicts a markedly worse prognosis compared to those who achieve a robust hematologic improvement (protocol 90-H-0146).

The current limitations of IST in SAA are: 1) the majority of the responses observed following initial h-ATG/CsA are partial with only a few patients achieving normal blood counts; 2) 1/3 of patients are refractory to initial h-ATG/CsA; 3) hematologic relapses occur in 35 percent of responders following initial response to h-ATG/CsA; 4) among relapsed patients chronic use of CsA is not infrequent which often leads to toxicities from the long term exposure to this drug (especially in older patients); 5) and clonal evolution is still observed in 10-15 percent of patients. Efforts to improve initial IST in treatment-naive patients with the addition of mycophenolate mofetil and sirolimus to standard h-ATG/CsA or use of lymphocytotoxic agents such as r-ATG/CsA or alemtuzumab have not yielded the expected better outcomes when compared to standard h-ATG/CsA (protocols 00-H-0032, 03-H-0193, and 06-H-0034). Because the majority of SAA patients in the US and worldwide are treated with IST due to lack of an human leukocyte antigen (HLA)-matched donor or inaccessibility to transplant, novel regimens are needed to overcome the current limitations of IST in SAA. Towards the goal of addressing these limitations we are proposing a regimen of cyclophosphamide (Cy) plus low dose CsA.

Cy has been proposed by the investigators at Johns Hopkins as an alternative IST regimen to h-ATG/CsA. In a pilot study, high dose Cy (200 mg/kg) yielded similar results to that observed for h-ATG/CsA. In a randomized study, at National Institute of Heart, Lung, and BIood (NHLBI), comparing high dose Cy (200 mg/kg) and h-ATG/CsA in treatment-na(SqrRoot) ve patients (protocol 97-H-0117), excess toxicity and deaths from invasive fungal infections were observed in the Cy arm which led to the discontinuation of this regimen. Recently reported long-term results from Johns Hopkins of 44 treatment-naive patients who received high dose Cy (200 mg/kg) as sole therapy for SAA showed that a greater number of complete responses were observed with few instances of relapse and clonal evolution noted with Cy when compared to h-ATG/CsA (historical comparison). In an accompanying editorial, the incidence of invasive fungal infections in this cohort were highlighted. Of note, antifungal prophylaxis against Aspergillus sp, the deadliest culprit when neutropenia is severe and prolonged, was not employed in the Hopkins high dose Cy protocol. In the Chinese experience, data presented in a recent meeting in Japan showed that lower doses of Cy (120 mg/kg) plus CsA achieved similar results reported by the Hopkins investigators with reduced toxicity. These data suggest that Cy has activity in SAA and could be a viable alternative to standard h-ATG/CsA if the immediate toxicities associated to prolonged neutropenia could be overcome.

In recent years we have observed a marked improvement in survival in our SAA patients especially among those who are non-responders to IST where pancytopenia remain persistent for months. A detailed analysis (shown in Section 2.4 Scientific and Clinical Justification of Protocol) showed that better antifungal supportive care in recent years contributed to a reduction of infection-related mortality in the months following IST among non-responders, who remain persistently neutropenic. This observation suggests that nowadays patients can be better supported through periods of neutropenia due to improved antifungal supportive care with agents that are better tolerated (compared to deoxycholate amphotericin B), retain a broad-spectrum of activity (especially against Aspergillus sp), and can be administered orally as an outpatient.

The fact that about one-third of initial refractory patients respond to retreatment and that late complications (relapse and clonal evolution) occur in about 40-50 percent of cases suggest that initial IST with h-ATG/CsA has important limitations. Therefore, we propose to investigate Cy + CsA as initial therapy in SAA. Our intention is not to recapitulate the high dose Cy regimen initially proposed by Hopkins (200 mg/kg) but instead, investigate lower doses proposed by the Chinese (120 mg/kg) in addition to low dose CsA (target therapeutic level 100 200 microg/L). The ability to better support patients during periods of neutropenia with better antifungals should allow for the immediate toxicity to be overcome and assess the activity of Cy in SAA.

The main objective of this study is to assess the safety and efficacy of Cy 120 mg/kg + low dose CsA (100 200 microg/L) in treatment-naive SAA. The primary endpoint will be hematologic response, defined as no longer meeting criteria for SAA, at 6 months. Secondary endpoints are relapse, robustness of hematologic recovery at 6 months, response at 3 months and 12 months, survival, clonal evolution to paroxysmal nocturnal hemoglobinuria (PNH), myelodysplasia and acute leukemia. The primary endpoint will be changes in absolute neutrophil count, platelet count, and reticulocyte count at 6 months. Secondary endpoints will include time to relapse, changes in cytogenetics, and time to death.

ELIGIBILITY:
* INCLUSION CRITERIA:

Severe aplastic anemia characterized by:

Bone marrow cellularity less than 30 percent (excluding lymphocytes)

AND

At least two of the following:

Absolute neutrophil count less than 500/ microL

Platelet count less than 20,000/ microL

Absolute reticulocyte count less than 60,000/ microL

Age greater than or equal to 2 years old

Weight greater than or equal to 12 kg

EXCLUSION CRITERIA:

Diagnosis of Fanconi anemia

Cardiac ejection fraction less than 30 percent (evaluated by ECHO)

Evidence of a clonal hematologic bone marrow disorder on cytogenetics. Patients with the presence of trisomy 8, loss of Y or del(20q) will not be excluded in the absence of dysplastic changes in the marrow. Patients with very severe neutropenia (ANC less than 200 /microL) will not be excluded initially if cytogenetics are not available or pending. If evidence of a clonal disorder is later identified, the patient will go off study.

Prior immunosuppressive therapy with high dose Cy or ATG

Infection not adequately controlled with appropriate therapy

Serologic evidence of HIV infection

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 30 days is likely

Subjects with cancer who are not considered cured, are on active chemotherapeutic treatment or who take drugs with hematological effects

Current pregnancy or unwillingness to take oral contraceptives or refrain from pregnancy if of childbearing potential

Not able to understand the investigational nature of the study or to give informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Townsley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenfeld S, Follmann D, Nunez O, Young NS. Antithymocyte globulin and cyclosporine for severe aplastic anemia: association between hematologic response and long-term outcome. JAMA. 2003 Mar 5;289(9):1130-5. doi: 10.1001/jama.289.9.1130. PMID 12622583
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Scheinberg P, Nunez O, Wu C, Young NS. Treatment of severe aplastic anaemia with combined immunosuppression: anti-thymocyte globulin, ciclosporin and mycophenolate mofetil. Br J Haematol. 2006 Jun;133(6):606-11. doi: 10.1111/j.1365-2141.2006.06085.x. PMID 16704434
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- [Derived] Scheinberg P, Townsley D, Dumitriu B, Scheinberg P, Weinstein B, Daphtary M, Rios O, Wu CO, Young NS. Moderate-dose cyclophosphamide for severe aplastic anemia has significant toxicity and does not prevent relapse and clonal evolution. Blood. 2014 Oct 30;124(18):2820-3. doi: 10.1182/blood-2014-05-573642. Epub 2014 Sep 3. PMID 25185712
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-H-0176.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAA Hematologic Response
Started | 22
Completed | 21
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | SAA Hematologic Response
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 16
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Blood Counts and Adverse Event Profile After 6 Months of Treatment.
Description: The safety endpoint will be toxicity profile after 6 months of treatment. The efficacy endpoint is complete response rate at 6 months, with complete response defined as blood counts no longer meeting the standard criteria for severe pancytopenia in severe aplastic anemia.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | SAA Hematologic Response
Number analyzed (Participants) | 21
participants
  Complete response | 4
  Partial Response | 5
  No Response | 12

ADVERSE EVENTS:
Arm/Group | SAA Hematologic Response
Serious Adverse Events (participants affected / at risk) | 16/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAA Hematologic Response (N=22)
Catheter-related infection (Infections and infestations) | 4 (4)
Bacterial infection (Infections and infestations) | 6 (6)
Fungal infection (Immune system disorders) | 3 (3)
Pnuemonia (Infections and infestations) | 7 (7)
Febril neutropenia (Blood and lymphatic system disorders) | 8 (8)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Lung abscess (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — perirectal abscess
sinus infection (Infections and infestations) | 1 (1)
petechiae (Blood and lymphatic system disorders) | 1 (1) — periorbital hemorrhage
blood infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes